CLINICAL TRIAL: NCT04510389
Title: Impact of Whey Protein Supplementation on Body Composition, Energy Expenditure and Biochemical Parameters of Patients Submitted to Bariatric Surgery
Brief Title: Impact of Whey Protein Supplementation on Body Weight and Metabolic Parameters of Bariatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Jacqueline Isaura Alvarez Leite, Full Professor, Federal University of Minas Gerais
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JLeite
Record Dates: First submitted 2019-01-18; First posted 2020-08-12 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Bariatric Surgery; Sarcopenia
Keywords: obesity; sarcopenia; bariatric surgery; protein
MeSH Terms: conditions — Sarcopenia; Obesity | interventions — maltodextrin; Whey

STUDY DESIGN:
Intervention Model Description: randomized
Who Masked: Participant, Investigator
Masking Description: Patient will receive indistinguishable sachets containing 30g of maltodextrin (placebo) or 30g whey protein. The sachets codification and patient allocation will be prepared by an individual without any contact with patients or the team which will follow patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): volunteers will receive 28 sachets containing 30g of maltodextrin to be consumed daily for 4 weeks. After that they will return to the 4-week visit and assessment when they will receive 28 sachets for the next 28 days when will return for the final vist and assessment.
  Interventions: Dietary Supplement: Maltodextrin
- Whey (Experimental): volunteers will receive 28 sachets containing 30g of whey protein to be consumed daily for 4 weeks. After that they will return to the 4-week visit and assessment when they will receive 28 sachets for the next 28 days when will return for the final vist and assessment.
  Interventions: Dietary Supplement: Whey

INTERVENTIONS:
Dietary Supplement: Maltodextrin — Bariatric patients with or without sarcopenia receiving maltodextrin
  Arms: Placebo
Dietary Supplement: Whey — Bariatric patients with or without sarcopenia receiving whey protein
  Arms: Whey

SUMMARY:
Obesity is a metabolic disorder, characterized by an increase in the body's fat mass, which will reflect an increase in total body weight. In Brazil, overweight accounts for 53.8% of the population, and of these 18.9% are obese. Surgical treatment is currently the most successful method for weight loss in patients with Grade III obesity and reduced associated morbidities. The general objective is to evaluate genetic, inflammatory, and dietary factors that would influence weight loss and the appearance of protein deficiency or sarcopenia in patients undergoing bariatric surgery and to evaluate the effects of protein supplementation for 8 weeks after the 18th postoperative month in the parameters evaluated. The study has a randomized, placebo-controlled, double-masked model. The patients will be selected in two bariatric surgery services accredited by the Brazilian Health Unic System (SUS) in the city of Belo Horizonte, Brazil.

The project has already been approved by the Brazilian Ethics committee CONEP/UFMG by nº. 75415317.8.0000.5149. Patients of both sexes over 20 years of age will be included, attending the hospitals of the project with regular follow-up in the postoperative period. Data on anthropometry, body composition, muscle strength, energy expenditure, and inflammatory profile will be collected. The data will be correlated with the evaluation of the presence of genetic polymorphisms.

DETAILED DESCRIPTION:
Specific objectives:

It is also objective to evaluate:

* To observe the food consumption between 18 and 24 months of surgery with respect to protein and caloric intake;
* Evolution of weight loss, lean mass, fat mass and metabolic rate before and after supplementation with WP or placebo;
* Changes in protein status (assessed by muscle strength and serum levels of total protein, albumin, prealbumin, ferritin, hemoglobin) before and after supplementation with WP or placebo
* The inflammatory blood profile (assessed by cytokine levels and before and after supplementation with WP or placebo).
* The influence of the rS9939609 polymorphism of the FTO gene on the nutritional status, biochemical and inflammatory parameters in the postoperative (after 18 months) of surgery;

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over 20 years of age
* Patients with regular follow-up in the postoperative period.

Exclusion Criteria:

* Patients with debilitating chronic diseases
* Severe vomiting
* Submitted to other surgical procedures before 18 months of surgery
* Patient with prostheses
* Use or introduction of drugs immunosuppressants or affecting metabolism

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Body Weight variation | 8th week
  measured in scale presented in kg
Muscle mass | 8th week
  measure by portable US

SECONDARY OUTCOMES:
Body Weight variation | 4th week
  measured in scale presented in kg
Resting metabolic rate | 4th week
  measured by indirect calorimetry in kcal/kg/day
Muscle mass | 4th week
  measure by portable US
SNP (FTO) detection | 1st week
  measure by polymerase chain reaction (PCR) in present or absence of A and T allele
Serum albumin | 4th week
  measured in serum in g/dL
Serum albumin | 8th week
  measured in serum in g/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratório de Aterosclerose e Bioquimica Nutricional, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No